CLINICAL TRIAL: NCT04821284
Title: Optimizing Ultrasound Enhanced Delivery of Therapeutics
Brief Title: Sonoporation and Chemotherapy for the Treatment of Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Flemming Forsberg (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Flemming Forsberg, Professor - Radiology, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20F.1207; R01CA199646 (NIH); JT 15477 (Other: JeffTrial Number)
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Oxaliplatin; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (sonazoid, ultrasound, chemotherapy) (Experimental): Patients receive standard of care chemotherapy consisting of gemcitabine hydrochloride and nab-paclitaxel IV over 60 minutes on days 1, 8 and 15 OR FOLFIRINOX IV on days 1 and 2. Treatments repeat every 28 days for up to 3 cycles for gemcitabine and nab-paclitaxel, and every 14 days for up to 7 cycles for FOLFIRINOX in the absence of disease progression or unacceptable toxicity. Patients also receive sonazoid IV over 20 minutes and undergo CEUS. Patients undergo CT or PET/CT or MRI during screening and as clinically indicated on study.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Nab-paclitaxel; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Other: Perflubutane Microbubble; Procedure: Contrast-Enhanced Ultrasound; Other: Quality-of-Life Assessment; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm II (chemotherapy) (Active Comparator): Patients receive standard of care chemotherapy consisting of gemcitabine hydrochloride and nab-paclitaxel IV over 60 minutes on days 1, 8 and 15 OR FOLFIRINOX IV on days 1 and 2. Treatments repeat every 28 days for up to 3 cycles for gemcitabine and nab-paclitaxel, and every 14 days for up to 7 cycles for FOLFIRINOX in the absence of disease progression or unacceptable toxicity. Patients undergo CT or PET/CT or MRI during screening and as clinically indicated on study.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Nab-paclitaxel; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Other: Quality-of-Life Assessment; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: 1-(2-Oxo-4-amino-1; 2-dihydropyrimidin-1-yl)-2-deoxy-2; 2-difluororibose, hydrochloride; 122111-03-9; 2'Deoxy-2'; 2'-Difluorocytidine; Hydrochloride; dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; nanoparticle paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; protein-bound paclitaxel
Drug: Fluorouracil — Given IV
  Other Names: 2,4-Dioxo-5-fluoropyrimidine; 5 Fluorouracil; 5 FU; 5 Fluorouracilum; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluoro-2,4(1H,3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU, 5-Fu; 51-21-8; 5FU; AccuSite; Carac; Fluoro Uracil; fluorouraci; Fluouracil; Flurablastin; Fluracedy; Fluracil; Fluril; Ribofluor; Ro 2-9757
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: 136572-09-3; Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
Drug: Leucovorin Calcium — Given IV
  Other Names: 1492-18-8; 5-Formyl Tetrahydrofolate; 5-Formyl-5,6,7,8-tetrahydrofolic Acid; 5-Formyl-5,6,7,8-tetrahydropteroyl-L-glutamic Acid; Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calcium N-(p-((((6RS)-2-amino-5-formyl-5,6,7,8-tetrahydro-4-hydroxy-6-pteridinyl)methyl)amino)benzoyl)-L-glutamate (1:1); Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor; Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; N-[4-[[(2-Amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amnio]benzoyl]-L-glutamic Acid; Calcium Salt (1:1); N-[p-[[(2-Amino-5-formyl-5,6,7,8-tetrahydro-4-hydroxy-6-pteridinyl)methyl]amino]benzoyl]glutamic Acid; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; 61825-94-3; [(1R,-2R)-1,2-cyclohexanediamine-N,N'][oxalato (2--)-O,O']platinum; [SP-4-2-(1R-trans)]-(1,2,cyclohexanediamine-N; N')[ethanedioato(2--)-O; O']platinum; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; oxalato (1R,2R-cyclohexanediamine)platinum(II); Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669; trans-l DACH oxalatoplatinum; trans-l diaminocyclohexane oxalatoplatinum
Other: Perflubutane Microbubble — Oxaliplatin
  Arms: Arm I (sonazoid, ultrasound, chemotherapy)
Procedure: Contrast-Enhanced Ultrasound — Undergo CEUS
  Arms: Arm I (sonazoid, ultrasound, chemotherapy)
Other: Quality-of-Life Assessment — Ancillary studies
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This phase I/II trial studies the effect of sonoporation in addition to standard of care chemotherapy in treating patients with pancreatic cancer. Sonoporation is a novel method that uses ultrasound and microbubbles to increase therapeutic effect by increasing uptake or enhance sensitization. Sonoporation together with chemotherapy may work better in treating patients with pancreatic cancer compared to chemotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and therapeutic efficacy of sonoporation on pancreatic ductal adenocarcinoma (PDAC) standard of care (SoC) treatment based on local progression-free and overall survival with the main endpoint being an increase in median progression-free survival of subjects by 8.7 months in the sonoporation group relative to controls.

SECONDARY OBJECTIVES:

I. To evaluate the effect of sonoporation on the median time to treatment failure (TTF) (in percent).

II. To evaluate the effect of sonoporation on the number of chemotherapy cycles subjects can undergo.

III. To evaluate the effect of sonoporation on tumor volume measured by clinical diagnostic ultrasound.

IV. To evaluate the effect of sonoporation on tumor perfusion using contrast enhanced ultrasound (CEUS) - specifically harmonic imaging (HI) and subharmonic imaging (SHI).

V. To evaluate the effect of sonoporation on tumor interstitial fluid pressures using subharmonic aided pressure estimation (SHAPE).

VI. To evaluate the effect of sonoporation on tumor volume using clinical diagnostic computed tomography (CT).

VII. To evaluate the effect of sonoporation on tumor stiffness using clinical ultrasound shear wave elastography (SWE).

VIII. To evaluate the effect of sonoporation on serum CA 19-9 concentrations. IX. Clinical benefit response, which is a measure of clinical improvement based on analgesic consumption, Eastern Cooperative Oncology Group (ECOG) performance status, and weight change.

X. To evaluate the effect of sonoporation on patient quality of life.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care chemotherapy consisting of gemcitabine hydrochloride and nab-paclitaxel intravenously (IV) over 60 minutes on days 1, 8 and 15 OR fluorouracil, irinotecan hydrochloride, leucovorin calcium and oxaliplatin (FOLFIRINOX) IV on days 1 and 2. Treatments repeat every 28 days for up to 3 cycles for gemcitabine and nab-paclitaxel, and every 14 days for up to 7 cycles for FOLFIRINOX in the absence of disease progression or unacceptable toxicity. Patients also receive sonazoid IV over 20 minutes and undergo CEUS. Patients undergo computed tomography (CT) or positron emission tomography (PET)/CT or magnetic resonance imaging (MRI) during screening and as clinically indicated on study.

ARM II: Patients receive standard of care chemotherapy consisting of gemcitabine hydrochloride and nab-paclitaxel IV over 60 minutes on days 1, 8 and 15 OR FOLFIRINOX IV on days 1 and 2. Treatments repeat every 28 days for up to 3 cycles for gemcitabine and nab-paclitaxel, and every 14 days for up to 7 cycles for FOLFIRINOX in the absence of disease progression or unacceptable toxicity. Patients undergo CT or PET/CT or MRI during screening and as clinically indicated on study.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years old
* Patient has a new diagnosis of PDAC and is scheduled to undergo SoC chemotherapy

  * (International Classification of Diseases [ICD]-10 C25.0 Malignant neoplasm: Head of pancreas, C25.1: Malignant neoplasm: Body of pancreas, C25.2 Malignant neoplasm: Tail of pancreas, C25.3 Malignant neoplasm: Pancreatic duct and C25.9 Malignant neoplasm: Pancreas, unspecified). Any ICD-10 code in the C25 section (malignant neoplasm of pancreas) will be acceptable
  * Histologically verified, locally advanced (stage II/III) or metastatic (stage IV) adenocarcinoma of the pancreas
* The PDAC must be visible on grayscale ultrasound prior to injection of ultrasound contrast
* Must be ambulatory with an ECOG performance status between 0 and 2
* Female patients of child-bearing potential must have a negative urine pregnancy test and use (and agree to continue to use throughout the study) one of the following forms of contraception from the screening Visit until completion of the first study follow-up visit: hormonal (oral, implant or injection) begun > 15 days prior to the screening visit, barrier (e.g., condom, diaphragm with spermicide), intra-uterine device or vasectomized partner (6 months minimum). Male patients must also agree to practice throughout the study an approved method of birth control.

  * (Note: To be considered NOT of child-bearing potential, female patients must be postmenopausal [with amenorrhea for at least 2 years prior to study entry] or surgically sterile [bilateral tubal ligation at least 6 months prior to study entry, or of a hysterectomy and/or bilateral oophorectomy])
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Conference on Harmonization (ICH)/Good Clinical Practice (GCP), and national/local regulations

Exclusion Criteria:

* Patient participated in an investigational study within 7 days prior to study entry (or, if longer, within five half-lives of the last dose of any investigational drug
* Patient has severe chronic obstructive pulmonary disease, or pulmonary hypertension or unstable cardiopulmonary conditions
* Patients who are medically unstable. For example:

  * Patients on life support or in a critical care unit
  * Patients with unstable occlusive disease (e.g., crescendo angina)
  * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia
  * Patients with uncontrolled congestive heart failure (New York Heart Association [NYHA] class IV)
  * Patients with recent cerebral hemorrhage
  * Patients who have undergone surgery within 24 hours prior to the study sonographic examination
* Patient with a history of any psychiatric disorder or cognitive impairment that would interfere with participation in the study in the opinion of the investigator
* Patient requires dialysis or has severely impaired renal function, defined as a serum creatinine >= 1.5 x ULN or calculated creatinine clearance < 45 mL/min at the screening visit
* Patient has severe impairment of liver function, defined as a serum albumin level =< 25 g/L and/or a prothrombin time international normalized ratio (INR) > 2.3 (or activated partial thromboplastin time [APTT] > 6 seconds above the upper limit of normal), or a Child Pugh Score C at the screening visit
* Patients diagnosed with human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV)
* Patients with a history of anaphylactic allergy to eggs or egg products, manifested by one or more of the following symptoms: generalized urticaria, difficulty in breathing, swelling of the mouth and throat, hypotension, or shock. (Subjects with non anaphylactic allergies to eggs or egg products may be enrolled in the study, but must be watched carefully for 1 hour following the administration of Sonazoid)
* Patients that are allergic to any other component of Sonazoid
* Any reason why, in the opinion of the investigator, the patient should not participate
* Patient is pregnant or is breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 3 years
  Gehan-Breslow-Wilcoxon test and Log-rank (Mantel-Cox) test will be used to compare progression free survival (PSF) between the groups with and without sonoporation.

SECONDARY OUTCOMES:
Number of chemotherapy cycles a subject can tolerate | Up to 3 years
  Gehan-Breslow-Wilcoxon test and Log-rank (Mantel-Cox) test will be used to compare number of chemotherapy cycles between the groups with and without sonoporation.
Overall survival | Up to 3 years
  Gehan-Breslow-Wilcoxon test and Log-rank (Mantel-Cox) test will be used to compare overall survival (PSF) between the groups with and without sonoporation.
Tumor volume changes | Up to 3 years
  Relative changes will be measured with ultrasound, computed tomography and/or magnetic resonance imaging and will also be compared between the groups with and without sonoporation.
Contrast enhanced ultrasound data | Up to 3 years
  Will provide perfusion and pressure estimates, which will be compared (individually and jointly) to subject outcomes in the groups with and without sonoporation as determined by the medical oncology team.
Tumor stiffness | Up to 3 years
  Will be measured as shear wave velocity obtained by ultrasound shear wave elastography and will be compared between the groups with and without sonoporation.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Thomas Jefferson University
Locations (2):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Adler O, Machado P, Vu T, Forsberg F, Gilja OH, Adam D. Perfusion Assessment in CEUS Imaging for Estimating Pancreatic Cancer Response to Sonoporation-Enhanced Chemotherapy. Ultrason Imaging. 2026 Jan;48(1):36-52. doi: 10.1177/01617346251367758. Epub 2025 Oct 24. PMID 41133726